CLINICAL TRIAL: NCT02902484
Title: A Phase 1b and Pharmacodynamic Study of Nintedanib Monotherapy for Advanced Pancreatic Cancer
Brief Title: Study of Nintedanib and Chemotherapy for Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to futility and lack of future funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Boehringer Ingelheim (Industry); The University of Texas Health Science Center at San Antonio (Other); South Plains Oncology Consortium (Network)
Responsible Party: Principal Investigator, Salwan Al Mutar MD MS, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 022016-083
Record Dates: First submitted 2016-09-02; First posted 2016-09-15 (Estimated); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nintedanib Monotherapy (Experimental): One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150, 200 mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib Monotherapy Followed by Combination Therapy of Nintedanib and Gemcitabine Plus nab-Paclitaxel
  Other Names: Ofev, Vargatef

SUMMARY:
The study will perform a clinical study evaluating the safety and tolerability of nintedanib when combined with standard chemotherapy (Gemcitabine + nab-Paclitaxel) for metastatic pancreatic cancer. It will utilize advanced imaging correlates including dynamic contrast enhanced Magnetic Resonance Imaging (DCE-MRI) which correlates with tumor grade and microvessel density.

DETAILED DESCRIPTION:
Preclinical data suggest nintedanib inhibits primary tumor growth in in vivo xenograft models of pancreatic cancer, as well as inhibiting metastasis in pancreatic cancer models. This effect appears primarily due to nintedanib anti-angiogenic properties. The study will perform a clinical study evaluating the safety and tolerability of nintedanib when combined with standard chemotherapy (Gemcitabine + nab-Paclitaxel) for metastatic pancreatic cancer. It will utilize advanced imaging correlates including dynamic contrast enhanced Magnetic Resonance Imaging (DCE-MRI) which correlates with tumor grade and microvessel density.

For each patient, treatment will have two phases: nintedanib monotherapy for a two week period (Days 1-14) followed by combination phase of nintedanib plus chemotherapy (Cycle 2+).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent prior to admission to the study;
2. Histologically or cytologically confirmed metastatic or locally advanced adenocarcinoma of the pancreas;
3. At least one measurable disease lesion according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1);
4. Age ≥ 18 years;
5. No more than one prior line of non-gemcitabine/nab-paclitaxel containing systemic therapy for metastatic/locally advanced pancreatic cancer;
6. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1;
7. Women of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration; (Note: contraception in patients with reproductive capacity will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least two years.)
8. Adequate biological parameters at baseline (obtained within 14 days prior to registration).
9. If elevated liver function tests develop at the time of initial presentation or develop during workup and are the result of mechanical obstruction of the biliary drainage by tumor compression or invasion, a biliary drain may be placed. If drainage allows the liver function tests to come within inclusion criteria, the patient may be enrolled.

Exclusion Criteria:

1. More than one systemic therapy regimen of any type for metastatic or locally advanced disease. Adjuvant gemcitabine that ended more than 6 months from diagnosis of recurrent disease is not considered as a regimen;
2. Prior treatment with nintedanib or any other VEGFR inhibitor;
3. Known hypersensitivity to nintedanib, gemcitabine and nab-Paclitaxal peanut or soya or any other trial drug, their excipients or to contrast media;
4. Chemo-, hormon-, radio-(except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug;
5. Radiotherapy to the target lesion within the past 3 months prior to baseline imaging
6. Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy;
7. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomization);
8. Leptomeningeal disease;
9. Radiographic evidence of cavitary or necrotic tumors;
10. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial;
11. Therapeutic anticoagulation with drugs requiring INR monitoring (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day);
12. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period;
13. History of clinically significant hemorrhagic or thromboembolic event in the past 6 months;
14. Known inherited predisposition to bleeding or thrombosis;
15. Significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion);
16. Proteinuria CTCAE grade 2 or greater;
17. Creatinine > 1.5 x ULN or GFR < 45 mL/min;
18. Hepatic function: total bilirubin outside of normal limits; ALT or AST > 1.5 ULN in pts without liver metastasis. For Pts with liver metastasis: total bilirubin outside of normal limits, ALT or AST > 2.5 ULN;
19. Coagulation parameters: International Normalized Ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN;
20. Absolute neutrophil count (ANC) < 1500/mL, platelets < 100,000/mL, Hemoglobin < 9.0 g/dl;
21. Any known active cancer other than pancreatic primary;
22. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy;
23. Active or chronic hepatitis C and/or B infection;
24. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug;
25. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study;
26. Pregnancy or breast feeding female;
27. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule;
28. Active alcohol or drug abuse;
29. Significant weight loss (> 20% of BW) within past 6 months prior to inclusion into the trial or actual body weight of less than 50 kg;
30. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectable, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salwan Al Mutar, MD, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 subjects were consented in which 1 subject withdrew consent and was not assigned to treatment.
Groups:
- Nintedanib 150 mg: One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150 mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
  Nintedanib: Nintedanib Monotherapy Followed by Combination Therapy of Nintedanib and Gemcitabine Plus nab-Paclitaxel
- Nintedanib 200 mg: One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 200 mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
  Nintedanib: Nintedanib Monotherapy Followed by Combination Therapy of Nintedanib and Gemcitabine Plus nab-Paclitaxel
Period: Nintedanib Monotherapy 150 mg
Arm/Group | Nintedanib 150 mg | Nintedanib 200 mg
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Nintedanib Monotherapy 200 mg
Arm/Group | Nintedanib 150 mg | Nintedanib 200 mg
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0
Period: Nintedanib 150 mg + Chemotherapy
Arm/Group | Nintedanib 150 mg | Nintedanib 200 mg
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Nintedanib 200 mg + Chemotherapy
Arm/Group | Nintedanib 150 mg | Nintedanib 200 mg
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nintedanib 150mg: One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150 mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
  Nintedanib: Nintedanib Monotherapy Followed by Combination Therapy of Nintedanib and Gemcitabine Plus nab-Paclitaxel
- Nintedanib 200mg: One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 200 mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
- Total: Total of all reporting groups
Arm/Group | Nintedanib 150mg | Nintedanib 200mg | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Continuous [Median (Full Range); unit: years] | 65 [58 to 74] | 63 [50 to 73] | 63 [50 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 10 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 9 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: A standard 3+3 phase 1 trial design will be used for Nintedanib monotherapy for a two week period (Days 1-14) followed by combination therapy of nintedanib plus chemotherapy. Two dose levels of nintedanib will be explored 150 mg BID and 200 mg BID. The combination phase will include gemcitabine + nab-paclitaxel, and nintedanib. Treatment will be administered intravenously on days 1, 8, 15 every 28 days.
  One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150 mg PO BID and 200mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
  MTD assessed after combination therapy.
Time Frame: Each 28 day cycle for up to 2 years
Measure: Number; unit: mg
Groups:
- All Participants: Two dose levels of nintedanib will be explored 150 mg BID and 200 mg BID. The combination phase will include gemcitabine + nab-paclitaxel, and nintedanib. Treatment will be administered intravenously on days 1, 8, 15 every 28 days.
  One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150 mg PO BID and 200mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
Arm/Group | All Participants
Number analyzed (Participants) | 13
mg | 200

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 3 years, 1 month.
Groups:
- Nintedanib 150 mg: One cycle of Nintedanib monotherapy followed by a total of eight cycles of both Nintedanib and the chemotherapeutic agents, or until disease progression, whichever comes first.
  1. Nintedanib dose escalation: 150mg PO BID
  2. Nab-paclitaxel: 125 mg/m2 day 1,8,15 every 28 days
  3. Gemcitabine: 1000 mg /m2 day 1,8,15 every 28 days
Arm/Group | Nintedanib 150 mg | Nintedanib 200 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib 150 mg (N=3) | Nintedanib 200 mg (N=10)
Neutropenia (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib 150 mg (N=3) | Nintedanib 200 mg (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (7)
Abscess of gluteal lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (5)
Azotemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (28) | 3 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Weightloss (Investigations) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burning sensation leg and head (General disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
chills (General disorders) | 1 (2) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Chronic Kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Consipation (Gastrointestinal disorders) | 0 (0) | 3 (5)
Creatinine increased (Investigations) | 1 (2) | 0 (0)
Creatinine decreased (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 6 (11)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Edema Face (General disorders) | 1 (1) | 0 (0)
Edema limbs (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated (Transamineses, AST/ALT, bilirubn) (Investigations) | 2 (5) | 3 (5)
enlarged prostate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (5) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
General weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (4)
Hairloss (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hip/Spine Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hyperuncemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 4 (8)
hypothyroid (Endocrine disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Itchy Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
vomiting (Gastrointestinal disorders) | 1 (4) | 3 (3)
Body Pain (General disorders) | 1 (2) | 6 (8)
Leg swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 7 (9)
Leukopenia (Metabolism and nutrition disorders) | 3 (61) | 2 (4)
neuropathy (Nervous system disorders) | 1 (1) | 8 (9)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Frequent Urination (Renal and urinary disorders) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Nasal congestion / drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Lymphocytopenia (Vascular disorders) | 3 (53) | 3 (7)
lower extremity cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 3 (27) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (30) | 3 (8)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Tingling in finger tips left hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (51) | 3 (3)
Oral Sensitivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Worsening of gluteal lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
nail infection (Infections and infestations) | 0 (0) | 1 (1)
Rash on back of head, arms and groin area (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pale colored stool (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02902484/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02902484/ICF_003.pdf